CLINICAL TRIAL: NCT07121959
Title: An Open-Label, Phase 1 Study to Characterize the Effects of Belzutifan on the Pharmacokinetics of a MATE1/2K Substrate, Metformin, in Healthy Adult Participants
Brief Title: A Study of Belzutifan (MK-6482) and Metformin in Healthy Adult Participants (MK-6482-039)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6482-039; MK-6482-039 (Other: MSD)
Record Dates: First submitted 2025-08-12; First posted 2025-08-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): On Day 1 of Period 1, a single dose of metformin will be administered.
  Interventions: Drug: Metformin
- Belzutifan with Metformin (Experimental): In Period 2, belzutifan will be administered every day for 5 consecutive days with a single dose of metformin coadministered on Day 4.
  Interventions: Drug: Metformin; Drug: Belzutifan

INTERVENTIONS:
Drug: Metformin — Oral Tablet
  Other Names: Metformin HCl
Drug: Belzutifan — Oral Tablet
  Other Names: MK-6482
  Arms: Belzutifan with Metformin

SUMMARY:
The goal of this study is to learn how belzutifan (MK-6482) affects the levels of metformin in a healthy person's body over time. Researchers will study levels of metformin in the blood and urine in healthy volunteers after taking metformin alone (Period 1) and metformin with belzutifan (Period 2).

ELIGIBILITY:
The main inclusion criteria include, but are not limited to:

* Is a continuous non-smoker for at least 3 months prior to dosing
* Has body mass index (BMI) ≥ 18.0 and ≤ 42.0 kg/m2
* Is able to swallow multiple tablets

The main exclusion criteria include, but are not limited to:

* Has a history of cancer (malignancy)
* Has a history of anemia within the last 5 years
* Has a known history or presence of metabolic acidosis, ketoacidosis, or lactic acidosis
* Has a hemoglobin level below the lower limit of normal
* Has a pulse oximetry reading less than 92% at rest
* Is known to be a cytochrome P450 (CYP2C19) poor metabolizer or likely poor metabolizer based on genotyping prior to the screening visit or is determined to be a CYP2C19 poor metabolizer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) for Metformin in Plasma | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Blood samples will be collected to determine the AUC0-inf of metformin in plasma.

SECONDARY OUTCOMES:
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 4 weeks
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants Who Discontinue Study Drug Due to an AE | Up to approximately 2 weeks
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Area Under the Concentration Versus Time Curve from 0 to the Last Quantifiable Sample (AUC0-last) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the AUC0-last of metformin.
Area Under the Concentration Versus Time Curve from 0 to 24 hours (AUC0-24) of Metformin | At designated timepoints (up to approximately 24 hours post-dose metformin)
  Plasma samples will be collected to determine the AUC0-24 of metformin.
Maximum Observed Concentration (Cmax) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the Cmax of metformin.
Plasma Drug Concentration of Metformin at Hour 24 (C24) | 24 hours post-dose metformin
  Plasma samples will be collected to determine the C24 of metformin.
Time to Maximum Concentration (Tmax) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the Tmax of metformin.
Apparent Terminal Half-life (t1/2) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the t1/2 of metformin.
Apparent Clearance (CL/F) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the CL/F of metformin.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Plasma samples will be collected to determine the Vz/F of metformin.
Total Amount of Metformin Excreted Unchanged in the Urine | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Urine samples will be collected to determine the total amount of metformin excreted unchanged in the urine.
Percentage of Metformin Excreted Unchanged in Urine | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Urine samples will be collected to determine the percentage of metformin excreted unchanged in urine.
Renal Clearance of Metformin | At designated timepoints (up to approximately 48 hours post-dose metformin)
  Urine samples will be collected to determine the renal clearance of metformin.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/